CLINICAL TRIAL: NCT01135381
Title: E-Coaching: IVR-Enhanced Care Transition Support for Complex Patients
Brief Title: IVR-Enhanced Care Transition Support for Complex Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of California, San Francisco (Other); US Department of Veterans Affairs (U.S. Federal Agency); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Christine Ritchie, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R18HS017786 (AHRQ)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Congestive Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: care transitions; information technology
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CHF patients, IVR-Enhanced Care (Experimental): Patients with congestive heart failure (CHF) who receive the interactive voice response (IVR) intervention.
  Interventions: Behavioral: IVR-Enhanced Care
- COPD patients, IVR-Enhanced Care (Experimental): Patients with chronic obstructive pulmonary disease (COPD) who receive the interactive voice response (IVR) intervention.
  Interventions: Behavioral: IVR-Enhanced Care
- CHF patients, Usual Discharge Care (No Intervention): Patients with congestive heart failure (CHF) who receive usual discharge care (no intervention).
- COPD patients, Usual Discharge Care (No Intervention): Patients with chronic obstructive pulmonary disease (COPD) who receive usual discharge care (no intervention).

INTERVENTIONS:
Behavioral: IVR-Enhanced Care — Those randomized to e-Coach will receive initial coaching in the hospital and then will be called by the interactive voice response-supported (IVR) system at specified intervals after discharge for monitoring. Any red flags noted through the IVR monitoring system will be transmitted to the care transition coaches, who contact patients and coach them on how to address problems identified.
  Other Names: e-Coach; IVR; IVRS; IVR Care Transition Support; Interactive voice response-supported system
  Arms: CHF patients, IVR-Enhanced Care; COPD patients, IVR-Enhanced Care

SUMMARY:
For complex medical patients, the transition from hospital to home-based care is a vulnerable period, placing the patient at high risk for adverse events. Using a Care Transition conceptual model, the investigators propose developing and evaluating, through a randomized controlled trial, "e-Coach," an Interactive-Voice-Response-supported (IVR) Care Transition coaching intervention, focused initially on patients hospitalized with heart failure or obstructive lung disease. This trial will test the primary hypothesis that the proportion of patients with one or more re-hospitalizations during a 90-day post-discharge follow-up period will be less in an IVRsupported care transition intervention (e-Coach) compared to a "usual care" comparison group.

DETAILED DESCRIPTION:
For complex medical patients, the transition from hospital to home-based care is a vulnerable period, placing the patient at high risk for adverse events, including the experience of a medical error or loss of community tenure. Recent successful studies have used a Care Transition Intervention (CTI), using a nurse who conducts home visits, telephone follow-up, and provides assistance at and after discharge. Although successful, this model is costly and and not feasible in settings serving geographically dispersed populations. We propose a cost-efficient technological solution to the problems presented by the traditional CTI through "e-Coach," an Interactive-Voice-Response-supported (IVR) Care Transition coaching intervention. We propose to develop and evaluate "e-Coach," by performing a randomized controlled trial of this intervention versus a usual care comparison group. Our Specific Aims are to: 1) Randomize 720 patients at high risk of transition-related errors (complex adult patients discharged alive after a hospitalization with congestive heart failure (CHF) or chronic obstructive pulmonary disease (COPD), from a geographically diverse area including many rural areas across Alabama and the South) to an IVR-supported care transition program ("e-Coach") versus a usual care comparison group. The IVR system will actively call patients at multiple intervals after discharge. In a stepped-care approach, the IVR will be further supported by a Care Transition nurse who monitors patient symptoms through the e-Coach IVR and supports patient self management through telephone-based interactions when needed, up to 3 months after discharge; 2) Evaluate use of the e-Coach by patients and healthcare providers; 3) Evaluate the impact of the e-Coach on patient outcomes, including 90 day rehospitalizations, successful community tenure over a 3 month period, medication discrepancies, and patient self-efficacy based on the previously validated Care Transition Measure; and 4) Quantify the cost associated with the e-Coach.

ELIGIBILITY:
Inclusion Criteria:

* CHF/COPD patients
* English-speaking
* Medicare beneficiaries

Amendment to Inclusion Criteria:

* Recruited non-Medicare eligible beneficiaries

Exclusion Criteria:

* Prognosis of 6 months or less
* Cognitive impairment with no available proxy/caregiver
* No possession of a phone

Amendments to exclusion criteria:

* heart or lung transplant recipients
* dialysis patients
* individuals already in the Cystic Fibrosis program or receiving intensive monitored care
* individuals with a ventricular assist device (LVAD; RVAD; BiVAD)
* individuals utilizing a pre-paid phone service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine S Ritchie, MD, MSPH, Principal Investigator — University of Alabama at Birmingham; Thomas K Houston, MD, MSPH, Study Director — University of Massachusetts, Worcester; Joshua Richman, MD, PhD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University Hospital and UAB Highlands, Birmingham, Alabama, United States

REFERENCES:
- [Background] Ritchie C, Richman J, Sobko H, Bodner E, Phillips B, Houston T. The E-coach transition support computer telephony implementation study: protocol of a randomized trial. Contemp Clin Trials. 2012 Nov;33(6):1172-9. doi: 10.1016/j.cct.2012.08.007. Epub 2012 Aug 19. PMID 22922245
- [Derived] Ritchie CS, Houston TK, Richman JS, Sobko HJ, Berner ES, Taylor BB, Salanitro AH, Locher JL. The E-Coach technology-assisted care transition system: a pragmatic randomized trial. Transl Behav Med. 2016 Sep;6(3):428-37. doi: 10.1007/s13142-016-0422-8. PMID 27339715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from multiple clinical units in a large tertiary care clinical facility in Alabama with a geographically wide, mostly rural catchment area.
  Recruitment period: 2/2010 to 3/2012.
Pre-assignment Details: 757 were discharged prior to completing their enrollment, and 304 did not meet other inclusion criteria. Thus, a total of 511 patients were enrolled and randomly assigned to groups.
Groups:
- CHF Patients, IVR-Enhanced Care: Patients with congestive heart failure (CHF) who receive the interactive voice response (IVR) intervention.
  IVR-Enhanced Care : Those randomized to e-Coach will receive initial coaching in the hospital and then will be called by the interactive voice response-supported (IVR) system at specified intervals after discharge for monitoring. Any red flags noted through the IVR monitoring system will be transmitted to the care transition coaches, who contact patients and coach them on how to address problems identified.
- COPD Patients, IVR-Enhanced Care: Patients with chronic obstructive pulmonary disease (COPD) who receive the interactive voice response (IVR) intervention.
  IVR-Enhanced Care : Those randomized to e-Coach will receive initial coaching in the hospital and then will be called by the interactive voice response-supported (IVR) system at specified intervals after discharge for monitoring. Any red flags noted through the IVR monitoring system will be transmitted to the care transition coaches, who contact patients and coach them on how to address problems identified.
Period: Overall Study
Arm/Group | CHF Patients, IVR-Enhanced Care | CHF Patients, Usual Discharge Care | COPD Patients, IVR-Enhanced Care | COPD Patients, Usual Discharge Care
Started | 189 | 185 | 69 | 68
Completed | 168 | 178 | 65 | 67
Not Completed | 21 | 7 | 4 | 1

BASELINE CHARACTERISTICS:
Population: A few patients were excluded from the final study groups. 6 patients died prior to discharge, 2 patients declined participation, and 4 patients became ineligible. After hospital discharge, 12 patients declined follow-up, we were unable to contact 5 for follow-up, and 4 became ineligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | CHF Patients, IVR-Enhanced Care | CHF Patients, Usual Discharge Care | COPD Patients, IVR-Enhanced Care | COPD Patients, Usual Discharge Care | Total
Number analyzed (Participants) | 168 | 178 | 65 | 67 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 94 | 89 | 33 | 38 | 254
  >=65 years | 74 | 89 | 32 | 29 | 224
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (12.5) | 63 (13.4) | 62 (13.4) | 61 (14.0) | 63 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 82 | 38 | 21 | 227
  Male | 82 | 96 | 27 | 46 | 251
Region of Enrollment [Number; unit: participants]
  United States | 168 | 178 | 65 | 67 | 478

OUTCOME MEASURES:

1. Primary Outcome: Re-hospitalizations
Time Frame: During the 30days after discharge
Measure: Number; unit: participants
Arm/Group | CHF Patients, IVR-Enhanced Care | CHF Patients, Usual Discharge Care | COPD Patients, IVR-Enhanced Care | COPD Patients, Usual Discharge Care
Number analyzed (Participants) | 168 | 178 | 65 | 67
participants | 27 | 26 | 8 | 14

2. Secondary Outcome: Rehospitalizations at 90 Days
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | CHF Patients, IVR-Enhanced Care | CHF Patients, Usual Discharge Care | COPD Patients, IVR-Enhanced Care | COPD Patients, Usual Discharge Care
Number analyzed (Participants) | 168 | 178 | 65 | 67
participants | 54 | 48 | 22 | 26

3. Secondary Outcome: Community Tenure
Description: The number of days a patient spends in the home versus the hospital at 30 days.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CHF Patients, IVR-Enhanced Care | CHF Patients, Usual Discharge Care | COPD Patients, IVR-Enhanced Care | COPD Patients, Usual Discharge Care
Number analyzed (Participants) | 168 | 178 | 65 | 67
days | 1.62 (4.6) | 1.48 (4.1) | 0.52 (1.8) | 1.6 (3.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period (2 years)
Description: There were no serious adverse events (SAE) or other adverse events as a result of the intervention. Any adverse events that occurred were expected outcomes, given the baseline health level of the participants.
Arm/Group | CHF Patients, IVR-Enhanced Care | CHF Patients, Usual Discharge Care | COPD Patients, IVR-Enhanced Care | COPD Patients, Usual Discharge Care
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/178 | 0/65 | 0/67
Other Adverse Events (participants affected / at risk) | 0/168 | 0/178 | 0/65 | 0/67

LIMITATIONS AND CAVEATS:
Limitations include generalizability. Our single healthcare system likely has unique characteristics. Readmission to the hospital is also a limited quality measure. There is currently no way to deem if readmissions are appropriate or avoidable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No